CLINICAL TRIAL: NCT05634096
Title: Oximetry for Diagnosis of Obstructive Sleep Apnea Syndrome in Children
Brief Title: Oximetry in Children for Sleep Apnea Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr. Iulia IOAN, Head of Pediatric Lung Function Department, Associate Professor, Central Hospital, Nancy, France
Other Study IDs: 2022PI161-318
Record Dates: First submitted 2022-11-22; First posted 2022-12-01 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep; Child; Polysomnography; Polygraphy
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Oximetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oximetry — Children underwent oximetry simultaneously with video-polygraphy or video-polysomnography in routine clinical practice. The data are retrospectively collected from the patient's recording.

SUMMARY:
Video-polygraphy or video-polysomnography (vP(S)G) is the reference exam for the diagnosis of obstructive sleep apnea syndrome (OSAS) in children as it allows the detection of the respiratory events presented by the child during sleep. This exam requires a one-night hospitalization and several sensors installed on the child's body, sometimes not well-accepted in children. Portable oximetry is an easier test to perform, better accepted by the child, and gives the desaturation index that may be used for the diagnosis of OSAS because most respiratory events are associated with desaturations. The hypothesis of this study is that the desaturation index obtained by the oximetry performed at the same time with the v(P(S)G) can identify a moderate-severe OSAS in children.

DETAILED DESCRIPTION:
Video-polysomnography (vPSG) with video surveillance and monitoring by a nurse to reposition the sensors if needed during the night is the gold standard exam for the diagnosis of obstructive sleep apnea syndrome (OSAS) in children. The vPSG gives the obstructive apnea-hypopnea index (OAHI), necessary for the diagnosis of OSAS and to determine its severity. But the vPSG is a rather cumbersome exam, sometimes difficult to perform in children, with several sensors and electrodes to install on a child's body (electroencephalogram (EEG), electromyogram (EMG), electrooculogram (EOG), nasal cannula, thoracoabdominal belts, pulse oximetry, body position) that is time-consuming for installation and analysis. Video-respiratory polygraphy (vPG) is very similar to vPSG but without EEG, EOG and EMG electrodes. vPG represents an alternative for the diagnosis of OSAS. However, these sleep examinations, vP(S)G, requires a number of electrodes and sensors to be installed on the child's body and one night of hospitalization.

The desaturation index obtained by simple portable oximetry could be used for the diagnosis of OSAS because most respiratory events are associated with desaturations. Portable oximetry is an easier test to perform. It is better accepted by the child because it only requires a finger or toe sensor and could be done on an outpatient basis or in the hospital.

The coupling of these 2 examinations, vP(S)G and oximetry, is part of our current routine practice. The hypothesis of this study is that the desaturation index obtained by the oximetry performed at the same time with the v(P(S)G) can identify an OSAS in children.

ELIGIBILITY:
Inclusion Criteria:

Children aged 2 to 18 years suspected of OSA who underwent a vP(S)G simultaneously with oximetry during the period June 2017 to June 2022.

Exclusion Criteria:

Children with non-interpretable recordings

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who underwent a vP(S)G simultaneously with oximetry during the period June 2017 to June 2022. Data of vP(S)G and of oximetry are retrospectively collected from the hospital recording of children who underwent these exams.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2023-01-02 (Estimated); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Desaturation index is different in moderate-severe OSAS | Baseline
  The number of desaturations per hour of recording obtained by oximetry between children with moderate-severe OSAS (defined as OAHI ≥ 5/h of sleep on the vP(S)G) and children without OSAS/with mild OSAS (defined as OAHI < 5/h of sleep )

SECONDARY OUTCOMES:
Sensitivity and specificity of desaturation index | Baseline
  Sensitivity and specificity of the number of desaturations per hour if recording obtained by oximetry alone for the identification of children with moderate-severe OSAS (defined as an OAHI ≥ 5 /h of sleep in vP(S)G).

CONTACTS AND LOCATIONS:
Overall Officials: Iulia IOAN, MD PhD, Principal Investigator — CHRU de Nancy
Locations (1):
- CHRU de Nancy, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Background] Kaditis A, Kheirandish-Gozal L, Gozal D. Pediatric OSAS: Oximetry can provide answers when polysomnography is not available. Sleep Med Rev. 2016 Jun;27:96-105. doi: 10.1016/j.smrv.2015.05.008. Epub 2015 Jun 4. PMID 26146027
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Sheldon SH, Spruyt K, Ward SD, Lehmann C, Shiffman RN; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):576-84. doi: 10.1542/peds.2012-1671. Epub 2012 Aug 27. PMID 22926173
- [Background] Van Eyck A, Lambrechts C, Vanheeswijck L, Van Hoorenbeeck K, Haentjens D, Boudewyns A, De Winter BY, Van Gaal L, De Backer W, Verhulst SL. The role of nocturnal pulse oximetry in the screening for obstructive sleep apnea in obese children and adolescents. Sleep Med. 2015 Nov;16(11):1409-1412. doi: 10.1016/j.sleep.2015.07.023. Epub 2015 Aug 18. PMID 26498244
- [Background] Trucco F, Rosenthal M, Bush A, Tan HL. The McGill score as a screening test for obstructive sleep disordered breathing in children with co-morbidities. Sleep Med. 2020 Apr;68:173-176. doi: 10.1016/j.sleep.2019.12.010. Epub 2019 Dec 28. PMID 32044554